CLINICAL TRIAL: NCT03701971
Title: Randomized Prospective Open-label Study Evaluating the Benefit of Music Therapy on Pruritus in Patients With Pruritic Dermatitis
Brief Title: Study Evaluating the Benefit of Music Therapy on Pruritus in Patients With Pruritic Dermatitis
Acronym: PRURI-MUSIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC18.0112
Record Dates: First submitted 2018-09-27; First posted 2018-10-10 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: evaluation of the benefit of music therapy on pruritus in patients with pruritic dermatitis compared to the application of an emollient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): * a medical examination
  * Before and after music therapy, patients will have to answer questionnaires :
  Before :
  Questionnaire 5D itch scale Itchy Quality of Life Pruritus assessment on the digital scale Questionnaire State-Trait Anxiety Inventory (STAI Y-A)
  After :
  Pruritus assessment on the digital scale Questionnaire State-Trait Anxiety Inventory (STAI Y-A) PGIC
  • Patients will then benefit from a balneotherapy session the next morning. Patients will have to answer questionnaires before and after balneotherapy :
  Before :
  Pruritus assessment on the digital scale Questionnaire State-Trait Anxiety Inventory (STAI Y-A)
  After :
  Pruritus assessment on the digital scale Questionnaire State-Trait Anxiety Inventory (STAI Y-A) PGIC
  Interventions: Other: evaluation of the intensity of pruritus
- Emollient cream (Active Comparator): * a medical examination
  * Before and after music therapy, patients will have to answer questionnaires :
  Before :
  * Questionnaire 5D itch scale
  * Itchy Quality of Life
  * Pruritus assessment on the digital scale
  * Questionnaire State-Trait Anxiety Inventory (STAI Y-A)
  After :
  * Pruritus assessment on the digital scale
  * Questionnaire State-Trait Anxiety Inventory (STAI Y-A)
  * PGIC
    * Patients will then benefit from a balneotherapy session the next morning. Patients will have to answer questionnaires before and after balneotherapy :
  Before :
  * Pruritus assessment on the digital scale
  * Questionnaire State-Trait Anxiety Inventory (STAI Y-A)
  After :
  * Pruritus assessment on the digital scale
  * Questionnaire State-Trait Anxiety Inventory (STAI Y-A)
  * PGIC
  Interventions: Other: evaluation of the intensity of pruritus

INTERVENTIONS:
Other: evaluation of the intensity of pruritus — evaluation of the intensity of pruritus with various questionnaires

SUMMARY:
Many clinical studies have shown the benefit of music therapy in various pathologies, including pain, and it is now established that the latter has a complementary therapeutic interest. Its most frequently identified indications are the fight against acute or chronic pains, the reduction of anxiety, depression and stress, as well as memory disorders such as Alzheimer's disease.

The main modes of action of music therapy involve sensory, cognitive, psychological and behavioral processes that are also found in pruritus.

Pruritus is defined as "an uncomfortable sensation causing the need to scratch. It has similarities with pain but also differences: relief by heat / cold, scratching / withdrawal behavior, localization on the skin, semi-mucous / ubiquitous ... etc.

The pathophysiology also has similarities, pruritus is born at the dermal-epidermal junction at the level of specific cutaneous receptors then follows the classical pathways through a 1st neuron, then the dorsal horn of the spinal cord and a second neuron. At the cerebral level, there is no single center of pruritus but several motor and sensory areas involved.

The similarities suggest that music therapy may have an interest in the management of chronic pruritus, especially since classical treatments (antihistamines, topical corticosteroids) have only partial efficacy in some dermatoses

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Patient with pruritic dermatosis whatever the etiology (psoriasis, atopic dermatitis, toxiderma, cutaneous lymphoma, chronic urticaria ...)
* Hospitalized in continuous hospitalization in the Dermatology Department
* Age of dermatosis ≥ 1 month
* Pruritus score ≥ 3/10 by numerical evaluation
* Patient having signed a consent form

Exclusion Criteria:

* Patient under the age of 18
* Major impairment of hearing function
* Presence of major cognitive disorders
* Refusal to participate
* Pregnant or lactating women
* Institutionalized or emergency patients
* Patient under legal protection regime
* Patient not affiliated to the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Variation in the intensity of pruritus | Hour 0 / Hour 1
  Variation in the intensity of pruritus on the digital scale of pruritus

SECONDARY OUTCOMES:
To study the effect of music therapy on the patient's anxiety | Hour 0 / Hour 1
  Completion of questionnaire State-Trait Anxiety Inventory (STAI Y-A)
To study the effect of music therapy according to the etiology of pruritus | Hour 0
  Completion of Questionnaire 5D itch scale
To study the impact of pruritic dermatitis on the quality of life of the patient | Hour 0
  Completion of Questionnaire Itchy Quality of Life
To study the satisfaction of the patients concerning the music session | Hour 1
  Completion of questionnaire PGIC (Patient's Global Impression of Change)

CONTACTS AND LOCATIONS:
Locations (1):
- Brest University Hospital, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning after result publication and ending fifteen years following the study completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Nowak D, Yeung J. Diagnostic et traitement du prurit. Can Fam Physician. 2017 Dec;63(12):925-931. French. PMID 29237631
- [Background] Leibovici V, Magora F, Cohen S, Ingber A. Effects of virtual reality immersion and audiovisual distraction techniques for patients with pruritus. Pain Res Manag. 2009 Jul-Aug;14(4):283-6. doi: 10.1155/2009/178751. PMID 19714267
- [Background] Elmariah SB, Lerner EA. Topical therapies for pruritus. Semin Cutan Med Surg. 2011 Jun;30(2):118-26. doi: 10.1016/j.sder.2011.04.008. PMID 21767774
- [Background] Misery L. [Pruritus: considerable progress in pathophysiology]. Med Sci (Paris). 2014 Dec;30(12):1123-8. doi: 10.1051/medsci/20143012015. Epub 2014 Dec 24. French. PMID 25537042
- [Background] Rossetti A, Chadha M, Torres BN, Lee JK, Hylton D, Loewy JV, Harrison LB. The Impact of Music Therapy on Anxiety in Cancer Patients Undergoing Simulation for Radiation Therapy. Int J Radiat Oncol Biol Phys. 2017 Sep 1;99(1):103-110. doi: 10.1016/j.ijrobp.2017.05.003. Epub 2017 May 8. PMID 28816136
- [Background] Hartling L, Newton AS, Liang Y, Jou H, Hewson K, Klassen TP, Curtis S. Music to reduce pain and distress in the pediatric emergency department: a randomized clinical trial. JAMA Pediatr. 2013 Sep;167(9):826-35. doi: 10.1001/jamapediatrics.2013.200. PMID 23857075
- [Background] Gold C, Wigram T, Elefant C. Music therapy for autistic spectrum disorder. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004381. doi: 10.1002/14651858.CD004381.pub2. PMID 16625601
- [Background] Vink AC, Birks JS, Bruinsma MS, Scholten RJ. Music therapy for people with dementia. Cochrane Database Syst Rev. 2004;(3):CD003477. doi: 10.1002/14651858.CD003477.pub2. PMID 15266489
- [Background] Cepeda MS, Carr DB, Lau J, Alvarez H. Music for pain relief. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004843. doi: 10.1002/14651858.CD004843.pub2. PMID 16625614
- [Background] Good M, Anderson GC, Ahn S, Cong X, Stanton-Hicks M. Relaxation and music reduce pain following intestinal surgery. Res Nurs Health. 2005 Jun;28(3):240-51. doi: 10.1002/nur.20076. PMID 15884029
- [Background] Good M, Picot BL, Salem SG, Chin CC, Picot SF, Lane D. Cultural differences in music chosen for pain relief. J Holist Nurs. 2000 Sep;18(3):245-60. doi: 10.1177/089801010001800306. PMID 11847812
- [Background] Burrai F, Micheluzzi V, Zito MP, Pietro G, Sisti D. Effects of live saxophone music on physiological parameters, pain, mood and itching levels in patients undergoing haemodialysis. J Ren Care. 2014 Dec;40(4):249-56. doi: 10.1111/jorc.12078. Epub 2014 Jul 1. PMID 24980265
- [Background] Gutgsell KJ, Schluchter M, Margevicius S, DeGolia PA, McLaughlin B, Harris M, Mecklenburg J, Wiencek C. Music therapy reduces pain in palliative care patients: a randomized controlled trial. J Pain Symptom Manage. 2013 May;45(5):822-31. doi: 10.1016/j.jpainsymman.2012.05.008. Epub 2012 Sep 24. PMID 23017609
- [Background] Kahloul M, Mhamdi S, Nakhli MS, Sfeyhi AN, Azzaza M, Chaouch A, Naija W. Effects of music therapy under general anesthesia in patients undergoing abdominal surgery. Libyan J Med. 2017 Dec;12(1):1260886. doi: 10.1080/19932820.2017.1260886. PMID 28452603
- [Background] Lesiuk T. The Effect of Mindfulness-Based Music Therapy on Attention and Mood in Women Receiving Adjuvant Chemotherapy for Breast Cancer: A Pilot Study. Oncol Nurs Forum. 2015 May;42(3):276-82. doi: 10.1188/15.ONF.276-282. PMID 25901379
- [Background] Hole J, Hirsch M, Ball E, Meads C. Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. Lancet. 2015 Oct 24;386(10004):1659-71. doi: 10.1016/S0140-6736(15)60169-6. Epub 2015 Aug 12. PMID 26277246
- [Background] Chen SJ, Xiao XL, Zhang L. The effect of music therapy on anxiety or depression status of severe male burn patients. J Chin Metallurgical Ind Med. 2005;3:328-329.
- [Background] Standley JM. Music research in medical/dental treatment: meta-analysis and clinical applications. J Music Ther. 1986 Summer;23(2):56-122. doi: 10.1093/jmt/23.2.56. PMID 10301218
- [Background] Hauck M, Metzner S, Rohlffs F, Lorenz J, Engel AK. The influence of music and music therapy on pain-induced neuronal oscillations measured by magnetencephalography. Pain. 2013 Apr;154(4):539-547. doi: 10.1016/j.pain.2012.12.016. Epub 2012 Dec 28. PMID 23414577
- [Background] Kordovan S, Preissler P, Kamphausen A, Bokemeyer C, Oechsle K. Prospective Study on Music Therapy in Terminally Ill Cancer Patients during Specialized Inpatient Palliative Care. J Palliat Med. 2016 Apr;19(4):394-9. doi: 10.1089/jpm.2015.0384. Epub 2016 Feb 19. PMID 26894922
- [Background] Gallagher LM, Lagman R, Walsh D, Davis MP, Legrand SB. The clinical effects of music therapy in palliative medicine. Support Care Cancer. 2006 Aug;14(8):859-66. doi: 10.1007/s00520-005-0013-6. Epub 2006 Mar 15. PMID 16538499
- [Background] Choi S, Park SG, Bellan L, Lee HH, Chung SK. Crossover clinical trial of pain relief in cataract surgery. Int Ophthalmol. 2018 Jun;38(3):1027-1033. doi: 10.1007/s10792-017-0554-y. Epub 2017 Jun 20. PMID 28639089
- [Background] Hoareau SG, De Diego E, Guetin S. [Pain management and music therapy]. Rev Infirm. 2016 Jan;(217):31-3. doi: 10.1016/j.revinf.2015.10.025. French. PMID 26743370
- [Background] Bates D, Bolwell B, Majhail NS, Rybicki L, Yurch M, Abounader D, Kohuth J, Jarancik S, Koniarczyk H, McLellan L, Dabney J, Lawrence C, Gallagher L, Kalaycio M, Sobecks R, Dean R, Hill B, Pohlman B, Hamilton BK, Gerds AT, Jagadeesh D, Liu HD. Music Therapy for Symptom Management After Autologous Stem Cell Transplantation: Results From a Randomized Study. Biol Blood Marrow Transplant. 2017 Sep;23(9):1567-1572. doi: 10.1016/j.bbmt.2017.05.015. Epub 2017 May 19. PMID 28533058
- [Background] Tarikci N, Kocaturk E, Gungor S, Topal IO, Can PU, Singer R. Pruritus in Systemic Diseases: A Review of Etiological Factors and New Treatment Modalities. ScientificWorldJournal. 2015;2015:803752. doi: 10.1155/2015/803752. Epub 2015 Jul 9. PMID 26240837
- [Background] Hon KL, Pong NH, Wang SS, Lee VW, Luk NM, Leung TF. Acceptability and efficacy of an emollient containing ceramide-precursor lipids and moisturizing factors for atopic dermatitis in pediatric patients. Drugs R D. 2013 Mar;13(1):37-42. doi: 10.1007/s40268-013-0004-x. PMID 23456759
- [Background] Hon KL, Kung JSC, Ng WGG, Leung TF. Emollient treatment of atopic dermatitis: latest evidence and clinical considerations. Drugs Context. 2018 Apr 17;7:212530. doi: 10.7573/dic.212530. eCollection 2018. PMID 29692852
- [Background] Jacobi A, Mayer A, Augustin M. Keratolytics and emollients and their role in the therapy of psoriasis: a systematic review. Dermatol Ther (Heidelb). 2015 Mar;5(1):1-18. doi: 10.1007/s13555-015-0068-3. Epub 2015 Jan 21. PMID 25604924
- [Background] Seccareccia D, Gebara N. Pruritus in palliative care: Getting up to scratch. Can Fam Physician. 2011 Sep;57(9):1010-3, e316-9. No abstract available. PMID 21918143
- [Background] Goutos I, Clarke M, Upson C, Richardson PM, Ghosh SJ. Review of therapeutic agents for burns pruritus and protocols for management in adult and paediatric patients using the GRADE classification. Indian J Plast Surg. 2010 Sep;43(Suppl):S51-62. doi: 10.4103/0970-0358.70721. PMID 21321658
- [Background] Moncrieff G, Cork M, Lawton S, Kokiet S, Daly C, Clark C. Use of emollients in dry-skin conditions: consensus statement. Clin Exp Dermatol. 2013 Apr;38(3):231-8; quiz 238. doi: 10.1111/ced.12104. PMID 23517354
- [Background] Misery L. Itch Management: General Principles. Curr Probl Dermatol. 2016;50:35-9. doi: 10.1159/000446039. Epub 2016 Aug 23. PMID 27578069
- [Background] Takeuchi S, Oba J, Esaki H, Furue M. Pruritus of patients with atopic dermatitis in daily life and their experience of therapeutic effects: results of a web-based questionnaire survey. Br J Dermatol. 2015 Jul;173(1):250-2. doi: 10.1111/bjd.13557. Epub 2015 Mar 27. No abstract available. PMID 25421804
- [Background] Weisshaar E, Szepietowski JC, Darsow U, Misery L, Wallengren J, Mettang T, Gieler U, Lotti T, Lambert J, Maisel P, Streit M, Greaves MW, Carmichael AJ, Tschachler E, Ring J, Stander S. European guideline on chronic pruritus. Acta Derm Venereol. 2012 Sep;92(5):563-81. doi: 10.2340/00015555-1400. No abstract available. PMID 22790094
- [Derived] Demirtas S, Houssais C, Tanniou J, Misery L, Brenaut E. Effectiveness of a music intervention on pruritus: an open randomized prospective study. J Eur Acad Dermatol Venereol. 2020 Jun;34(6):1280-1285. doi: 10.1111/jdv.16149. Epub 2020 Jan 14. PMID 31838780